CLINICAL TRIAL: NCT01503658
Title: Clinical Trial to Evaluate the Influence of Genotype of Drug Metabolizing Enzyme or Transporter and Drug-drug Interactions on the Pharmacokinetics/Pharmacodynamics of Clopidogrel in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate the Influence of Genotype on the Pharmacokinetics/Pharmacodynamics of Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Professor, Seoul National University Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGX_Clopidogrel_001
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Influence of Genotype of Drug Metabolizing Enzyme or Transporter on the Pharmacokinetics/Pharmacodynamics of Clopidogrel; Influence of Aspirin on the Pharmacokinetics/Pharmacodynamics of Clopidogrel
Keywords: Clopidogrel,; Aspirin,; Pharmacogenomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clopidogrel+Aspirin (Experimental): Clopidogrel on Day 1, Aspirin on Day 2 - Day 14, Clopidogrel + Aspirin Day 15, Aspirin on Day 16 - Day 28, Clopidogrel + Aspirin Day 29
  Interventions: Drug: Clopidogrel+Aspirin

INTERVENTIONS:
Drug: Clopidogrel+Aspirin — Clopidogrel 75 mg, Aspirin 100 mg

SUMMARY:
This study has an open-label, five-period, single-sequence design. The purpose of this study is as follows;

1. Primary

   * To evaluate the influence of genotype of drug metabolizing enzyme or transporter on the pharmacokinetics/pharmacodynamics of clopidogrel
   * To evaluate the influence of aspirin on the pharmacokinetics/pharmacodynamics of clopidogrel
2. Secondary

   * To explore the representative biomarkers for the variable pharmacokinetics/pharmacodynamics of clopidogrel
   * To evaluate the influence of genotype of drug metabolizing enzyme or transporter on the drug-drug interactions between aspirin and clopidogrel
   * To explore the representative biomarkers for the drug-drug interactions between aspirin and clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male subjects aged 20 - 45 years.
* 2. A body weight in the range of 50 kg (inclusive) - 90 kg (exclusive) and a body mass index (BMI) in the range 18.5 kg/m2 (inclusive) - 27 kg/m2 (inclusive).
* 3. Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully. informed about the study procedures.

Exclusion Criteria:

* 1. Presence or history of hypersensitivity or allergic reactions to drugs including investigational product (clopidogrel or aspirin)
* 2. Clinically relevant abnormal medical history that could interfere with the objectives of the study.
* 3. A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug.
* 4. A subject whose lab test results are as follows; Platelet count or PT, aPTT < 0.9 x lower limit of reference range of > 1.1 x upper limit of reference range.
* 5. A subject whose SBP is over 160 mmHg or below 90 mmHg and DBP is over 100 mmHg or below 50 mmHg.
* 6. Presence or history of drug abuse or positive result in urine drug screening test.
* 7. Participation in other clinical trial within 2 months before first dose.
* 8. Use of CYP inducer (ex. rifampin) within 4 weeks before first dose.
* 9. Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication or vitamin substances within 1 week before first dose.
* 10.Use of grapefruit juice within 1 week before first dose.
* 11. Blood donation during 2 months or apheresis during 1 month before the study.
* 12. Use of alcohol over 21 units/weeks
* 13. Smoking of more than 10 cigarettes/days within 3 months before first dose.
* 14. Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Clopidogrel | Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h postdose on Day 1, Day 15 and Day 29
  Plasma concentration of clopidogrel and active metabolite of clopidogrel
Pharmacodynamics of clopidogrel | Predose and 4, 24 h postdose on Day 1, Day 15 and Day 29
  Relative inhibition of platelet aggregation by aggregometer or VerifyNow

SECONDARY OUTCOMES:
mRNA/microRNA/endogenous metabolite | predose on Day 1, Day 8, Day 15, Day 22 and Day 29
  mRNA of PON1 and CYP2C19, CYP3A5, MDR1 microRNA endogenous metabolite

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea

REFERENCES:
- [Derived] Oh J, Shin D, Lim KS, Lee S, Jung KH, Chu K, Hong KS, Shin KH, Cho JY, Yoon SH, Ji SC, Yu KS, Lee H, Jang IJ. Aspirin decreases systemic exposure to clopidogrel through modulation of P-glycoprotein but does not alter its antithrombotic activity. Clin Pharmacol Ther. 2014 Jun;95(6):608-16. doi: 10.1038/clpt.2014.49. Epub 2014 Feb 24. PMID 24566733